CLINICAL TRIAL: NCT00718770
Title: Rexinoid Therapy for Poorly Differentiated Thyroid Cancer: A Pilot Clinical Trial and Correlation to Retinoid and PPARy Receptor Expression
Brief Title: A Pilot Clinical Trial for Poorly Differentiated Thyroid Cancer - Correlation to Retinoid and Peroxisome-proliferator-activated Receptor (PPARy) Expression
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: American Cancer Society, Inc. (Other); Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 07-0727.cc
Record Dates: First submitted 2008-07-17; First posted 2008-07-21 (Estimated); Results first posted 2014-01-17 (Estimated); Last update posted 2014-01-17 (Estimated); Status verified 2013-12

CONDITIONS: Thyroid Cancer
Keywords: Not respond; Radioactive iodine; Therapy; Shows signs; Aggressive behavior
MeSH Terms: conditions — Thyroid Neoplasms; Aggression | interventions — Bexarotene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Bexarotene (Experimental): Open label - all patients receive intervention
  Interventions: Drug: Bexarotene

INTERVENTIONS:
Drug: Bexarotene — Bexarotene will be given by mouth once a day every day for 1 year. The dose to be used will be 300 mg/m2.
  Other Names: LGD-1069

SUMMARY:
This study plans to learn more about a drug called bexarotene for the treatment of advanced thyroid cancer. Subjects are asked to be in this study because they have thyroid cancer that will not respond to radioactive iodine therapy and shows signs of aggressive behavior.

Bexarotene has been FDA approved for the treatment of a type of skin cancer called cutaneous T-cell lymphoma, but has not been FDA approved for this use. Bexarotene is investigational in the treatment of thyroid cancer.

The purpose of this research study is to test how well the study drug works in humans. The study doctors want to know if:

1. The subjects thyroid cancer gets smaller while you are taking the study drug.
2. The subjects thyroid cancer takes up radioactive iodine better after treatment with the study drug than before treatment.

ELIGIBILITY:
Inclusion Criteria:

* Subject must have a histologically/cytologically confirmed diagnosis of papillary, follicular, or anaplastic thyroid cancer (any follicular cell derived thyroid cancer).
* Subjects must have evidence of follicular cell-derived thyroid cancer progression. In patients with anatomically stable disease, PET positive lesions will also be eligible given the poor prognostic risk for PET positive thyroid cancer.
* Subjects must not be eligible for surgical resection.
* Subjects must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) criteria.
* Subjects must have laboratory values that fall within certain ranges.
* Subjects must be age 18 years or older.
* Subjects must provide written informed consent prior to any study procedures being performed.
* Females of childbearing potential must have a negative pregnancy test prior to enrollment.
* All eligible subjects must be willing to use adequate contraception throughout the duration of the study.
* Subjects must be willing to submit a primary tumor tissue sample for immunohistochemical analysis.
* Subjects have the option of providing one additional test tube of blood taken at baseline, 6 months and 1 year for banking of plasma for potential future studies (no genetic testing will be conducted). The current planned analysis is for the assessment of a potential peripheral marker for rexinoid responsive cancer - leukemia inhibitory factor (LIF)

Exclusion Criteria:

* Subjects with a known history of hyperlipidemia refractory to treatment.
* Subjects with a known history of hypertriglyceridemia refractory to treatment.
* Subjects with leukopenia below the reference range for the University of Colorado Hospital (UCH) laboratory.
* Subjects, who are pregnant, have a desire to become pregnant or are breastfeeding.
* Subjects who are unwilling or unable to comply with study medication administration, or study guidelines, as determined by the investigator.
* Subjects with any prior history of malignancy with the exception of adequately treated basal cell skin cancer, in situ cervical cancer or other cancer for which the subject has been disease free for 3 years or more.
* Subjects without radiographically assessable disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2008-11; Primary Completion 2013-01 (Actual); Study Completion 2013-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua Klopper, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Cancer Center, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients were recruited from a medical clinic from 01/15/2009 to 01/14/2010
Pre-assignment Details: The patients must fit all inclusion criteria and have had a 4 week washout from any systemic or radiation therapy. As an open-label, single arm trial, there was no group assignment. Patients were excluded only if they did not meet inclusion or had exclusion criteria
Groups:
- Bexarotene: Open label - all patients received the intervention
  Bexarotene : Bexarotene was given by mouth once a day every day for 1 year. The dose used was 300 mg/m2.
Period: Overall Study
Arm/Group | Bexarotene
Started | 10
Completed | 2
Not Completed | 8
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 1
Not completed — Lack of Efficacy | 1
Not completed — Adverse Event | 1

BASELINE CHARACTERISTICS:
Groups:
- Bexarotene: Open label - all patients receive intervention
  Bexarotene : Bexarotene will be given by mouth once a day every day for 1 year. The dose to be used will be 300 mg/m2.
Arm/Group | Bexarotene
Number analyzed (Participants) | 10
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 5
  >=65 years | 5
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.3 (8.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8
  Male | 2
Region of Enrollment [Number; unit: participants]
  United States | 10

OUTCOME MEASURES:

1. Primary Outcome: Change in Tumor Size
Description: To assess the tumor response of recurrent or metastatic radioiodine resistant thyroid cancer to bexarotene therapy using standard RECIST criteria
Time Frame: 1 year
Population: Adults with radioiodine resistant metastatic follicular cell derived thyroid cancer
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Bexarotene
Number analyzed (Participants) | 10
cm | 4.7 (0.2)

ADVERSE EVENTS:
Time Frame: 1 year
Arm/Group | Bexarotene
Serious Adverse Events (participants affected / at risk) | 0/10
Other Adverse Events (participants affected / at risk) | 4/10
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Bexarotene (N=10)
hyperlipidemia (Blood and lymphatic system disorders) | 4 (4)

LIMITATIONS AND CAVEATS:
Small numbers of participants with higher than expected numbers of patients not eligible and who could not complete trial due to lack of efficacy or drug side effects

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes